CLINICAL TRIAL: NCT06590194
Title: A Phase I/IIa, Open-label, Dose-escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Preliminary Anti-tumor Activity of PH009-1 in Patients With EGFR Mutation Locally Advanced or Metastatic NSCLC
Brief Title: PH009-1 in Patients With EGFR Mutation Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Puhe Pharmaceutical Technology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH009-101
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; EGFR; C797S
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 75mg, QD (Experimental): PH009-1 75mg QD orally administered, receive a single dose orally, followed by a 4-day washout period. Then, the same dose of PH009-1 will be administered QD, every 21 days a cycle until disease progression or not tolerated
  Interventions: Drug: PH009-1 tablet
- 150mg, QD (Experimental): PH009-1 150mg QD orally administered, receive a single dose orally, followed by a 4-day washout period. Then, the same dose of PH009-1 will be administered QD, every 21 days a cycle until disease progression or not tolerated
  Interventions: Drug: PH009-1 tablet
- 300mg, QD or 150mg, BID (Experimental): PH009-1 300mg QD or 150mg BID orally administered, receive a single dose orally, followed by a 4-day washout period. Then, the same dose of PH009-1 will be administered QD, every 21 days a cycle until disease progression or not tolerated
  Interventions: Drug: PH009-1 tablet
- 450mg, QD or 225mg, BID (Experimental): PH009-1 450mg QD or 225mg BID orally administered, receive a single dose orally, followed by a 4-day washout period. Then, the same dose of PH009-1 will be administered QD, every 21 days a cycle until disease progression or not tolerated
  Interventions: Drug: PH009-1 tablet
- 600mg, QD or 300mg, BID (Experimental): PH009-1 600mg QD or 300mg BID orally administered, receive a single dose orally, followed by a 4-day washout period. Then, the same dose of PH009-1 will be administered QD, every 21 days a cycle until disease progression or not tolerated
  Interventions: Drug: PH009-1 tablet
- 750mg, QD or 375mg, BID (Experimental): PH009-1 750mg QD or 375mg BID orally administered, receive a single dose orally, followed by a 4-day washout period. Then, the same dose of PH009-1 will be administered QD, every 21days a cycle until disease progression or not tolerated
  Interventions: Drug: PH009-1 tablet

INTERVENTIONS:
Drug: PH009-1 tablet — PH009-1 will be administered in fasting state
  Other Names: PH009-1

SUMMARY:
The study will contain three stages: Phase I includes dose escalation phase (i.e., phase Ia) and dose expansion phase (i.e., phase Ib). Once the dosage regimen is confirmed, the sponsor can decide to start the cohort expansion phase (i.e., phase IIa)

DETAILED DESCRIPTION:
phase Ia (Dose Escalation Phase) Approximately 17-96 subjects will be enrolled, dose escalation will be implemented by combining accelerated escalation with "3+3" design and safety evaluation requirements as specified. The total number of the subjects will depend upon the number of dose escalation necessary.

Phase Ib (Dose Expansion Phase): 2 to 3 doses selected from escalation doses, up to 20 subjects (subjects in dose escalation are involved) will be enrolled in each expansion arm, the total number of subjects will depend upon the number of dose expansions, expansions may adjusted depends upon the emerging data.

Phase IIa (Cohort Expansion): Approximately 20 subjects will be enrolled in each expansion cohort. Sample size may be adjusted based on emerging data.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, signed informed consent form before any trial-related processes.
2. Histological or cytological confirmed diagnosis of unresectable locally advanced or metastatic NSCLC.
3. Subjects must have NSCLC harboring one or more active EGFR mutations.
4. patients must have at least one measurable tumor lesion per RECIST v1.1 criteria as per Investigator's assessment.
5. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1.
6. Life expectancy ≥12 weeks.
7. Adequate hematologic and organ function per protocol.
8. WOCBP must have a negative serum and/or urine pregnancy test result within 7 days prior to the first dose of PH009-1.

Exclusion Criteria:

1. Treatment with any of the following:

   Prior treatment with an EGFR-TKI within 8 days prior to the first dose of PH009-1; Prior treatment with immunotherapy or biotherapy within 4 weeks prior to the first dose of PH009-1; Radiotherapy (palliative radiotherapy completed at least 2 weeks prior to the first dose of Ph009-1 can be enrolled) within 4 weeks prior to the first dose of PH009-1; Herbal therapy that has anti-tumor effects within 2 weeks prior to the first dose of PH009-1; Mitomycin and nitrosourea within 6 weeks prior to the first dose of PH009-1; Oral fluorouracil such as tegafur and capecitabine within 2 weeks prior to the first dose of PH009-1; Chemotherapy (except for mitomycin, nitrosourea, and fluorouracil oral drugs), or other anti-tumor drugs for the treatment of NSCLC within 4 weeks prior to the first dose of PH009-1. Marketed and/or experimental drug treatment for EGFR C797S mutations.
2. Is currently participating and receiving investigational therapy or using an investigational device, or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the investigational product, whichever is longer, prior to the first dose of PH009-1.
3. Is expected to require any other form of anti-tumor therapy while on study.
4. Unresolved toxicity greater than CTCAE v5.0 Grade 1 from prior anti-tumor therapy prior to the first dose.
5. Medical history of severe eye disease or skin disease without recovery to CTCAE v5.0 Grade 0 or 1 prior to the first dose.
6. Any of the following cardiovascular diseases within the last 6 months: include but not limited to QTc interval ≥ 470 msec.
7. Medical history of ILD.
8. Subjects with gastrointestinal disorders that may affect oral administration or interfere with the absorption of PH009-1, or severe gastrointestinal disease within 4 weeks prior to the first dose of PH009-1 and did not recover to ≤ CTCAE v5.0 Grade 2.
9. Major surgery or significant traumatic injury occurring within 4 weeks prior to the first dose of PH009-1 or anticipation of need for a major surgery during the study.
10. Has any bleeding tendency or coagulopathy within 6 months prior to the first dose of PH009-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose escalation and dose expansion: Incidence of dose-limiting toxicities (DLTs), Incidence and severity of treatment-emergent adverse events (TEAEs) with severity determined according to National Cancer Institute (NCI) CTCAE v5.0 | Up to approximately 2 years
  To evaluate the safety and tolerability of PH009-1 and to determine the maximal tolerable dose (MTD), or recommended phase II dose (RP2D).
Cohort expansion: Objective Response Rate (ORR) | Up to approximately 2 years
  To evaluate the preliminary anti-tumor activity at the selected dose(s) of oral PH009-1 according to RECIST v1.1.
Cohort expansion: Incidence and severity of AEs, with severity determined according to NCI CTCAE v5.0. | Up to approximately 2 years
  To evaluate the safety at the selected dose(s) of oral PH009-1.

SECONDARY OUTCOMES:
Peak plasma Concentration （Cmax） | Up to approximately 2 years
  To evaluate the pharmacokinetic (PK) characteristics of PH009-1 when given orally following single and multiple doses
Time to reach maximum concentration (Tmax) | Up to approximately 2 years
  To evaluate the pharmacokinetic (PK) characteristics of PH009-1 when given orally following single and multiple doses
Area under the plasma concentration versus time curve (AUC) | Up to approximately 2 years
  To evaluate the pharmacokinetic (PK) characteristics of PH009-1 when given orally following single and multiple doses
Disease Control Rate (DCR) | up to approximately 2 years
  To obtain a preliminary evaluation of the anti-tumor activity of PH009-1 according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Dose escalation and expansion: Objective Response Rate (ORR) | Up to approximately 2 years
  To obtain a preliminary evaluation of the anti-tumor activity of PH009-1 according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Duration of Reaponse (DOR) | up to approximately 2 years
  To obtain a preliminary evaluation of the anti-tumor activity of PH009-1 according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Progression-free survival (PFS) | up to approximately 2 years
  To obtain a preliminary evaluation of the anti-tumor activity of PH009-1 according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Time to progression (TTP) | up to approximately 2 years
  To obtain a preliminary evaluation of the anti-tumor activity of PH009-1 according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
overall survival (OS) | up to approximately 2 years
  To obtain a preliminary evaluation of the anti-tumor activity of PH009-1 according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
The concentration of PH009-1 in cerebrospinal fluid (CSF). | Up to approximately 2 years
  To characterise concentration of PH009-1 in CSF
The EGFR gene mutation status in circulating tumor deoxyribonucleic acid (ctDNA) | Up to approximately 2 years
  Confirm EGFR mutation status and evaluate the relationship between different EGFR mutations and drug responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdon, China

IPD SHARING:
Plan to Share IPD: No